CLINICAL TRIAL: NCT06896201
Title: Comfortage - Integration of Biomarkers, Genetic and Clinical Risk Factors for AD Prevention Strategies
Brief Title: Comfortage - AD Prevention Strategies
Acronym: Comfortage-P4
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 7334
Record Dates: First submitted 2025-02-26; First posted 2025-03-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer Disease; Subjective Cognitive Impairment; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Exercise Therapy; Nutritional Status

STUDY DESIGN:
Intervention Model Description: Interventional, cross-sectional, clinical trial without drug and without device
Masking Description: This study do not involve drug
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCD/MCI (Other): This 2 years study will include 100 individuals from two distinct clinical categories:
  * subjects with subjective cognitive decline
  * subjects with mild cognitive decline
  Interventions: Diagnostic Test: Neuropsychological Assessments and Other Questionnaires; Biological: Blood Exams, Fluid Biomarkers, Genetics; Other: Connectivity Analysis; Device: Physical Activity; Device: Healthentia; Device: Eligence; Other: Nutrition

INTERVENTIONS:
Diagnostic Test: Neuropsychological Assessments and Other Questionnaires — A brief assessment of the cognitive status will be performed by the means of Mini-Mental State Examination (MMSE), Clinical Dementia Rating Scale (CDR-SB), Activities of the Daily Living (ADL) and Instrumental Activities of the Daily Living (IADL) scales. Moreover, extended neuropsychological assessments assessing memory, language, executive functions, attention and visuospatial perception will be conducted by trained neuropsychologists, as per clinical practice. Concerning depression and behavioural / neuropsychiatric symptoms, which are known to be relevant in cognitive decline and ageing, data will be collected by the means of Neuropsychiatric Inventory (NPI). Additional questionnaires about subjective cognitive decline, quality of sleep (Pittsburgh scale) and cognitive reserve (CRIq) will be conducted on some subgroups of subjects.
Biological: Blood Exams, Fluid Biomarkers, Genetics — All patients will undergo a blood samples collection at T0 and T4, as per clinical practice. Additional blood samples will be collected stored and processed according to literature recommendation-based standardized operating procedures.. Blood will be collected into EDTA tubes and will be immediately refrigerated and centrifugated at 2000x g for 10 minutes. Plasma will then be aliquoted in 0.5 ml polypropylene vials and frozen at -80°C. Levels of blood biomarkers of amyloidopathy, tauopathy, neurodegeneration and neuroinflammation will be measured using the Lumipulse G assays (Fujirebio) and the Multiplex assays for Ella (Biotechne). Whole blood samples will be used for genetic analysis, which will include the determination of APOE genotype
Other: Connectivity Analysis — Functional Magnetic Resonance Imaging (fMRI) and/or high-density electroencephalography (EEG) will be used to assess connectivity in selected group of subjects. EEG data will be collected during four 5-minute runs of alternating eyes-open and eyes-closed conditions using a 128-electrode high-density EEG system.
  The EEG spectral coherence analysis will evaluate the functional coupling between the brain areas under study. Brain connectivity measures will be computed for each frequency band and for each subject, to be used as measure of weight of the graph in a graph analyses.
  A subsample of subjects will be also investigated with connectivity measures of MRI by applying FA e DTI technique. All the data will be collected both at baseline and after a 2-years-period during which the prevention and intervention strategies will be performed.
Device: Physical Activity — Participants will be proposed an unsupervised, monitored exercise program consisting of three 60-minute sessions of moderate-intensity aerobic exercise (40%-85% of their maximum heart rate) each week. To track exercise intensity. The activity will be personalized according to specific attitude of each subjects including walking session, bike sessions or swim sessions. The type, frequency and intensity of the activity will be recorded by means of a commercially available wearables (Garmin Vivosmart 4, Garmin Vivosmart 5) and the Healthentia application. Those non using the wearables will keep a diary of the activity. Study investigators will ensure both protocol adherence and participant safety through regular follow-up telephone contacts.
Device: Healthentia — Healthentia, developed by Innovation Sprint, is a Software as a Medical Device (SaMD) designed for remote patient monitoring, virtual coaching, and automatic alerts using real-world data. It has been successfully used in over 20 studies and integrates features like teleconsultations, activity tracking, medication management, and support for wearable devices. It provides a patient companion app, offering remote patient monitoring and self-reporting, personalized advice or content in the form of dialogues. It is designed to optimize and improve patient engagement and ensure data integrity. The software facilitates daily self-reporting, providing information to patients and collecting other current data through self-reported questionnaires (health status, physical activity, quality of life, etc.), which will be crucial in order to control the adherence of patients to the program
Device: Eligence — Based Platform exercising the brain and the cognitive skills through 35+ games and activities designed by specialized health experts. It offers over 30 games focusing on cognitive skills such as memory, reasoning, attention, orientation, executive functions, construction skills, and language. It allows healthcare professionals to create personalized training sessions, monitor performance in real-time, and generate detailed evaluation reports. Accessible from any device, it is aimed at individuals in early stages of dementia or rehabilitation phases. In our clinical study, subjects will be trained on seven cognitive programs, which can be executed at home with or without assistance and supervision of a Health Professional (who can easily create personalized sessions to follow-up at distance) and/or an informal carer
Other: Nutrition — Participants will follow a personalized nutrition plan, as per clinical practice, receiving dietary advice derived by the same scheme already used in the FINGER project on prevention. The plan focuses on balanced, nutrient-rich meals, based on the reduction of carbohydrate assumption and stable inclusion of seeds, vegetables, fish and omega 3 aliments in the diet that may protect the brain through anti-inflammatory and antioxidant properties. A diary of the meals will be recorded in a diary included in the Healthentia application. No integrated meals or nutraceutical product will be used.

SUMMARY:
Study is Interventional, cross-sectional, clinical trial without drug and without device

ELIGIBILITY:
Inclusion Criteria:

* subjective cognitive decline, defined as self-experienced persistent decline in cognitive capacity in comparison with a previously normal status and unrelated to an acute event; normal performance on standardised cognitive tests adjusted for age, sex, and education; decline cannot be explained by psychiatric or other neurologic disease, medical disorder, medication, or substance use; no functional impact on daily life activities
* mild cognitive decline, defined as persistent decline in cognitive performance (in comparison with a previous status) reported by the subject or by an informed caregiver; or observed by change on longitudinal cognitive testing; cognitive performance below expected range for that individual based on cognitive test performance (adjusted for age, sex, and education); performs daily life activities independently (but cognitive difficulty may result in detectable but minimal functional impact on the more complex activities of daily life, either self-reported or corroborated by a study partner); Clinical Dementia Rating Scale = 0.5
* Ability to sign and understand the informed consent form

Exclusion Criteria:

* Age under 50 or over 85 years
* Non-native Italian speakers
* Non degenerative and secondary forms of dementia
* Previous or current participation in clinical trials with anti-amyloid agents

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Changes in cognitive performance and quality of life through cognitive scales (MiniMental State Examination) | after 36 months
  Statistically significant differences in changes in cognitive performance and quality of life after a 2-year intervention period, stratified by clinical, genetic, connectivity, and/or biomarker profiles through cognitive scales as MiniMental State Examination.
Changes in cognitive performance and quality of life through cognitive scales (Clinical Dementia Rating Scale) | after 36 months
  Statistically significant differences in changes in cognitive performance and quality of life after a 2-year intervention period, stratified by clinical, genetic, connectivity, and/or biomarker profiles through cognitive scale as Clinical Dementia Rating Scale (CDR-SB).
Changes in cognitive performance and quality of life through cognitive scales (Activities of the Daily Living) | after 36 months
  Statistically significant differences in changes in cognitive performance and quality of life after a 2-year intervention period, stratified by clinical, genetic, connectivity, and/or biomarker profiles through cognitive scale as Activities of the Daily Living (ADL).
Changes in cognitive performance and quality of life through cognitive scales (Instrumental activities of the daily living) | after 36 months
  Statistically significant differences in changes in cognitive performance and quality of life after a 2-year intervention period, stratified by clinical, genetic, connectivity, and/or biomarker profiles through cognitive scale as Instrumental Activities of the Daily Living (IADL) scales.
Changes in cognitive performance and quality of life through questionnaires (Quality of sleep) | after 36 months
  Statistically significant differences in changes in cognitive performance and quality of life after a 2-year intervention period, stratified by clinical, genetic, connectivity, and/or biomarker profiles through questionnaire as the quality of sleep (Pittsburgh scale).
Changes in cognitive performance and quality of life through questionnaires (Cognitive reserve) | after 36 months
  Statistically significant differences in changes in cognitive performance and quality of life after a 2-year intervention period, stratified by clinical, genetic, connectivity, and/or biomarker profiles through questionnaires as the cognitive reserve (CRIq).

SECONDARY OUTCOMES:
Measure of improvement in cognitive functioning | after 36 months
  A greater than 20% improvement in cognitive functioning, as measured by standardized cognitive assessment tool as MiniMental State Examination, after a 2-year intervention period
Measure of improvement in cognitive functioning | after 36 months
  A greater than 20% improvement in cognitive functioning, as measured by standardized cognitive assessment tool as MontReal Cognitive Assessment (MOCA), after a 2-year intervention period
Measure of improvement in quality of life | after 36 months
  A greater than 35% improvement in quality of life, assessed through validated questionnaire as quality of sleep (Pittsburgh scale), following the 2-year intervention period
Measure of improvement in quality of life | after 36 months
  A greater than 35% improvement in quality of life, assessed through validated questionnaire as cognitive reserve (CRIq), following the 2-year intervention period
inflammatory blood biomarker levels | after 36 months
  Measurable and clinically relevant changes in AD neurodegenerative and inflammatory blood biomarker levels after the 2-year intervention period, correlating these changes with cognitive outcomes
Measure of improvement in user satisfaction | after 36 months
  A greater than 45% improvement in user satisfaction and interaction with the novel tools and interventions, as measured by satisfaction questionnaire , after the 2-year intervention period
Measure of changes in brain connectivity | after 36 months
  Measurable and clinically relevant changes in brain connectivity as resulted by electroencephalography (EEG) analyses after the 2-year intervention period, correlating these changes with cognitive outcomes.
  Regarding EEG analysis, data will be acquired during four successive 5-min runs of alternating eyes-open and eyes-closed conditions using a high-density EEG (128 cephalic electrodes). Frequency bands of interest will be delta (2-4 Hz), theta (4-8 Hz), alpha1 (8-10.5 Hz), alpha2 (10.5-13 Hz), beta1 (13-20 Hz), beta2 (20-30 Hz) and gamma (30-40 Hz).